CLINICAL TRIAL: NCT03297307
Title: Prospective: Mother and Child Health Outcomes After Maternal Bariatric Surgery
Brief Title: Mother and Child Health Outcomes After Maternal Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0821-17-EP
Record Dates: First submitted 2017-07-26; First posted 2017-09-29 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: This is a prospective intervention study of female bariatric surgical patients and their children. The dyads, consisting of one female bariatric patients and one child living in the home, will be enrolled in the study. Half of the children will attend the dietary, physical activity, and psychological counseling with the mother prior to her surgery, and the other half of the children will not receive the behavioral intervention. Outcomes from each mother-child dyad will be measured at baseline, and 3 and 6 months postoperatively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother-Child with Intervention (Experimental): Children will attend presurgical visits with their mother
  Interventions: Behavioral: Presurgical Counseling
- Mother-Child Non-Intervention (No Intervention): Children will not attend presurgical visits with their mother

INTERVENTIONS:
Behavioral: Presurgical Counseling — Children will attend the presurgical counseling visits with their mother
  Other Names: No Intervention
  Arms: Mother-Child with Intervention

SUMMARY:
Childhood obesity has been a growing problem with more than 30% of children between 6 and 19 years old being considered overweight or obese. Obese children are at increased risk of developing diabetes, heart disease, metabolic syndrome, and are susceptible to the sociological effects of being overweight. Obesity is a multifactorial disease, is often familial and multi-generational, and studies have shown that parental obesity can increase the risk of a child becoming obese. Currently, one of the most successful treatment options for obesity is bariatric surgery. The Nebraska Medicine Bariatric Center offers patients counseling in improved dietary management, methods to increase physical activity, and psychological support. As part of the programs standard-of-care, each bariatric surgical patient receives consultation with a dietician, psychologist, and an exercise physiologist. We propose that mothers who are enrolled in the surgical weight loss program bring their children to attend the presurgical specialist consultation. Subjects enrolled in the study will have their height, weight, and physical activity assessed at preoperative and postoperative study visits. Study subjects will also complete questionnaires of their self-reported physical activity and eating habits at these study visits. The goal of this pilot study is to examine whether this behavioral intervention will have an impact on the overall health and weight of children whose mothers have received bariatric surgery.

DETAILED DESCRIPTION:
This is a prospective intervention study of female bariatric surgical patients and their children. The dyads, consisting of one female bariatric patients and one child living in the home, will be enrolled in the study. Half of the children will attend the dietary, physical activity, and psychological counseling with the mother prior to her surgery, and the other half of the children will not receive the behavioral intervention. Outcomes from each mother-child dyad will be measured at baseline, and 3 and 6 months postoperatively (Visit BL-2, Visit PO-3, and Visit PO-6). The primary outcome measured from each dyad will be BMI, and secondary outcomes will be physical activity and energy expenditure (as measured by an accelerometer at each research study visit) and self-reported diet and physical activity (as measured by questionnaires completed at each research study visit).

Each bariatric surgical patient will receive a consultation with a dietician, psychologist, and an exercise physiologist as standard-of-care. These specialist consultations usually take place sequentially in the same day. The intervention aspect of this study is to include the child with the mother for these specialist consultations. The dietician will educate the patient as to dietary modifications that will be needed both before and after bariatric surgery. The psychologist will review any existing psychological conditions with the patient and discuss behavioral and pharmaceutical management of these conditions in conjunction with the bariatric surgery. The exercise physiologist will discuss physical restrictions to exercise and modifications to an exercise regimen that can be properly performed by the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-55 at the time of surgery
2. Consent to provide access to medical records for medical history
3. Will receive weight loss procedure (sleeve gastrectomy or gastric bypass) at Nebraska Medicine
4. Have children ages 8-17 (at the time of the mother's surgery) living in the home
5. Consent to wear an activity tracker device for 7 days after designated visits.

Exclusion Criteria:

1. Complication of bariatric procedure post-operatively that would significantly affect weight loss (extended period of TPN, clinically significant leak, major organ failure, severe protein malnutrition or failure to thrive)
2. Body contouring within the first year (panniculectomy, etc.).
3. Are pregnant or become pregnant during the study

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Maternal weight loss | presurgical, 3 mos, 6 mos
  Weight loss
Child weight loss | presurgical, 3 mos, 6 mos
  weight loss

SECONDARY OUTCOMES:
Maternal Activity level | presurgical, 3 mos, 6 mos
  activity level
Child Activity Level | presurgical, 3 mos, 6 mos
  activity level
Maternal diet | presurgical, 3 mos, 6 mos
  Self-reported diet
Child diet | presurgical, 3 mos, 6 mos
  self-reported diet

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Tanner, MD, Principal Investigator — UNMC
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be made available to other researchers